CLINICAL TRIAL: NCT02167867
Title: Evaluation of Efficacy, Usability and Labeling Comprehension for Over-the-Counter Use of the Erchonia Corporation ZERONA® Z6 for Body Contouring of the Waist, Hips and Thighs
Brief Title: Study of Over-The-Counter Use of Low Level Laser Light Therapy for Body Contouring of the Waist, Hips and Thighs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EC_Z6_OTC
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Circumference Reduction
Keywords: body contouring; circumference reduction; body shaping; low level laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lay End Users (Experimental): Employees of the test sites (that were fitness centers or spas) who were provided with a User's Manual to operate the ZERONA Z6 to administer 6 40-minute evenly spaced treatments over 2 consecutive weeks to the front and back of the waist, hips and thighs of one Treatment Subject.
  Interventions: Device: Treatment Subject Group
- Treatment Subject Group (Experimental): Treatment subjects received 6 40-minute evenly spaced treatments to the hips, waist and thighs (20 minutes to the front side and 20 minutes to the back side) with the ZERONA Z6 over 2 consecutive weeks. The ZERONA Z6 contains 6 17.25 milliWatts (mW) 635 nanometers (nm) laser diodes.
  Interventions: Device: Lay End Users

INTERVENTIONS:
Device: Lay End Users — Lay End Users administer 40 minutes of treatment with the ZERONA Z6 to the waist, hips and thighs (20 minutes to the front side and 20 minutes to the back side) of a Treatment Subject, 6 times evenly spaced across two consecutive weeks.
  Arms: Treatment Subject Group
Device: Treatment Subject Group — Treatment subject received 6 40-minute evenly spaced treatments to the hips, waist and thighs (20 minutes to the front side and 20 minutes to the back side) with the ZERONA Z6 over 2 consecutive weeks. The ZERONA Z6 contains 6 17.25 milliWatts (mW) 635 nanometers (nm) laser diodes.
  Arms: Lay End Users

SUMMARY:
The purpose of this study is to test the ability of the lay end user to understand the information contained in the User's Guide; to correctly identify patients who are suitably qualified to receive treatment; and to correctly administer the treatment with the Erchonia ZERONA® Z6 for circumference reduction of the waist, hips and thighs in an over-the-counter setting.

DETAILED DESCRIPTION:
The Erchonia ZERONA® Z6 is a low level laser light therapy device that has been approved by the United States Food and Drug Administration (FDA) for use by licensed medical professionals to help to reduce the circumference of the hips, waist and thighs.

This study is to see if the Erchonia ZERONA® Z6 can be used by lay (non-medical professional) people to treat others to help to reduce the circumference of the hips, waist and thighs.

ELIGIBILITY:
Lay End Users

Inclusion Criteria:

* 18 years of age or older
* Able to read and write English.
* Employees of the study test sites

Treatment Subjects

Inclusion Criteria

* 18 years of age or older
* Body Mass Index (BMI) <= 30 kg/m2

Exclusion Criteria

* Pregnancy
* Open wounds (sores, cuts, ulcers, etc.) on or around the waist, hips and/or thighs
* Currently have or are being treated for any cancerous growths on or around the waist, hips and/or thighs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zapolsky, Principal Investigator
Locations (1):
- Lifetime Fitness, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lay End Users: Employees of the test sites that were fitness centers or spas who were provided with a User's Manual to operate the ZERONA Z6 to administer 6 40-minute evenly spaced treatments over 2 consecutive weeks to the front and back of the waist, hips and thighs of a Treatment Subject.
- Treatment Subject Group: Subjects who received active treatments with the study device administered by the Lay End Users.
Period: Overall Study
Arm/Group | Lay End Users | Treatment Subject Group
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Subject Group: Treatment subjects received 6 40-minute evenly spaced treatments to the hips, waist and thighs (20 minutes to the front side and 20 minutes to the back side) with the ZERONA Z6 over 2 consecutive weeks. The ZERONA Z6 contains 6 17.25 milliWatts (mW) 635 nanometers (nm) light-emitting diodes.
- Total: Total of all reporting groups
Arm/Group | Lay End Users | Treatment Subject Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 22 | 42
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
Body Weight [Mean (Standard Deviation); unit: pounds] | NA (NA) — Measure of weight was not recorded to Lay End Users as it is not relevant to this group | 152.75 (25.59) | NA (NA) — Measure of weight was not recorded to Lay End Users as it is not relevant to this group; therefore, average values cannot be calculated.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | NA (NA) — Body Mass Index was not measures for Lay End Users as the measure is not relevant to this group. | 24.68 (2.06) | NA (NA) — Body Mass Index was not measures for Lay End Users as the measure is not relevant to this group; therefore average values cannot be calculated.

OUTCOME MEASURES:

1. Primary Outcome: Lay End User Ability to Correctly Choose Suitably Qualified Individuals to Get the ZERONA Z6 Treatments
Description: The number of lay end users who correctly evaluated and selected fully qualified individuals to get the ZERONA Z6 treatment was calculated.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Lay End Users: Employees of the test sites that were fitness centers or spas who were provided with a User's Manual to operate the ZERONA Z6 to administer 6 40-minute evenly spaced treatments over 2 consecutive weeks to the front and back of the waist. hips and thighs.
Arm/Group | Lay End Users
Number analyzed (Participants) | 22
participants | 22

2. Primary Outcome: Lay End User Ability to Correctly Use the ZERONA Z6 and Follow the Treatment Directions.
Description: The number of lay end users who correctly used the ZERONA Z6 to administer treatments by following the treatment administration protocol was calculated
Time Frame: two weeks
Measure: Number; unit: participants
Arm/Group | Lay End Users
Number analyzed (Participants) | 22
participants | 22

3. Primary Outcome: Average Change in Inches of Total Circumference Measurements for the Treatment Subject Group After 2 Weeks of Treatment With the ZERONA Z6
Description: Circumference in inches for the waist, hips and both thighs were measured and added together to give a total circumference measurement at baseline and at the end of the 2 weeks of treatment. The change in the total circumference measurement from baseline to the end of treatment was calculated. A decrease (-) in circumference measurement suggests study success and an increase (+) in circumference measurement suggests study failure. A decrease (-) of 3.52 inches (-3.52 inches) or more is positive for study success based on prior published results.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: inches
Groups:
- Treatment Subject Group: Individuals who got the active treatments with the ZERONA Z6.
Arm/Group | Treatment Subject Group
Number analyzed (Participants) | 22
inches | -3.72 (2.25)
Statistical Analysis 1: Comparison: Treatment Subject Group; t=+7.76; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- ZERONA Z6: ZERONA Z6 contains 6 17.25 milliWatts (mW) 635 nanometers (nm) light-emitting diodes. 6 40-minute evenly spaced treatments are administered over 2 consecutive weeks.
  ZERONA Z6: 20 minutes of treatment to the front side of the waist, hips and thighs and 20 minutes of treatment to the back side of the waist, hips and thighs.
Arm/Group | ZERONA Z6
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No